CLINICAL TRIAL: NCT00912769
Title: Outcome and Benefit After Total Knee Arthroplasty: Natural History of Muscle Power Recovery and Difference Between Different Surgical Approach
Brief Title: Knee Muscle Force Recovery After Minimally Invasive Surgery (MIS) Total Knee Replacement (TKR)
Acronym: MISTKR
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Dr. Chih-Hung Chang, Head of Division of Orthopedics, Far Eastern Memorial Hospital
Other Study IDs: 97025; 97025
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Total Knee Replacement Approach; Muscle Torque
Keywords: Total knee replacement; Subvastus; Midvastus; Isokinetic; Quadriceps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- subvastus approach/ midvastus approach: subvastus: vastus medialis oblique was not cut during operation midvastus: vastus medialis oblique was cut during operation
- Cybex: Knee extension/ flexion isometric and isokinetic performance of all cases were tested using Cybex

SUMMARY:
To compare muscle torque recovery between patients under subvastus approach and those under midvastus approach after total knee replacement

DETAILED DESCRIPTION:
Total knee Arthroplasty is a common operated surgery in each hospitals, and a lots of patients benefit from this surgery. Traditionally the frequently used surgical approach is parapatellar approach. However, recently the subvastus and midvastus approach has gained a world-wide population. These two methods had less damage to the quadriceps tendon and theoretically should have better post-operative muscle power recovery, less lateral retinaculum release because of better patellar tracking. The only differences between these two approaches are that the midvastus approach will split the vastus medialis muscle and denervation may occur. In this study we will use HSS or KSS functional score and Cybex dynamometer to evaluate the functional recovery, and use Merchant's view radiography to evaluate the result of patellar tracking. The follow-up period will not be limited and we will use mixed-model statistic's random effect to gain the natural history of muscle power recovery, which will become the base of other study. We can also compare the difference of results between PS type and CR type and different surgical approach. The natural history of the knee score will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients after subvastus approach or midvastus approach total knee replacement

Exclusion Criteria:

* patients with severe hypertension, heart disease or other problems which negatively influence the security of muscle test

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after total knee replacement without severe systemic disorders
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2003-10; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Pan-Ciao, Taipei, Taiwan